CLINICAL TRIAL: NCT04850209
Title: The Impact of Interactive Patient Education Based on WeChat Group on the Eradication Rate of Helicobacter Pylori
Brief Title: The Impact of WeChat Group Patient Education on the Eradication Rate of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021SDU-QILU-067
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Eradication; Patient Education
Keywords: helicobacter pylori; eradication; patient education; Wechat group

STUDY DESIGN:
Intervention Model Description: There are two randomized parallel groups in this study, control group and Wechat group.
Who Masked: Outcomes Assessor
Masking Description: The interventions are blind to follow-up personnel who collect and analyze compliance and the incidence of adverse events. The interventions are also blind to the UBT personnel.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Patients in this group will receive clarithromycin based bismuth-containing quadruple therapy, Vonoprazan fumarate 20 mg, colloidal bismuth pectin capsule 200 mg , amoxicillin 1000 mg and clarithromycin 500 mg, twice daily, 14 days.Patients will receive oral and written education
  Interventions: Other: oral and written education
- Wechat group (Experimental): Patients in this group will receive clarithromycin based bismuth-containing quadruple therapy, Vonoprazan fumarate 20 mg, colloidal bismuth pectin capsule 200 mg ,amoxicillin 1000 mg and clarithromycin 500 mg, twice daily, 14 days.Patients will receive oral and written education. And patients will be invited into a Wechat group to obtain interactive education through question and answer,which is provided by medical professionals.
  Interventions: Other: oral and written education; Other: Wechat group

INTERVENTIONS:
Other: oral and written education — oral and written education
Other: Wechat group — Wechat group: oral and written education plus Wechat group based interactive education provided by medical professional
  Arms: Wechat group

SUMMARY:
In this study, effects of oral and written education, WeChat education plus oral and written education on Helicobacter pylori eradication will be compared in a randomized way.

DETAILED DESCRIPTION:
There are two randomized parallel groups in this study, control group and Wechat group.All of the patients will be treated with Amoxicillin + Clarithromycin + Bismuth + Vonoprazan fumarate. In control group,the patients will be educated by oral and written way about the regimen. In Wechat group, the patients will be educated by Wechat oral and written way. Then, the eradication rates, compliance, adverse events, patients' satisfaction and experience will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 75 years old;
2. H. pylori infection confirmed by any two positive outcomes of rapid urease test (RUT), 13C-urea breath test (UBT) or histopathology.

Exclusion Criteria:

1. previous therapy for H. pylori;
2. with significant underlying disease (e.g. decompensated liver cirrhosis, renal failure or malignant tumors) that may interfere the study;
3. history of gastric surgery,
4. pregnancy or lactation;
5. the use of PPI or antibiotics during the 4 weeks prior to enrolment;
6. previous history of allergic reactions to any of the medications used in this protocol;
7. unable to use smartphone and wechat
8. unwilling or incapable to provide informed consents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
eradication rate in each group | 2 months
  Six weeks after completion of treatment，number of patients get H.pylori eradicated supported by negative 13C-UBT results will be investigated by an independent researcher.Then eradication rate in each group will be calculated by using intention-to-treat analysis and per-protocol analysis.

SECONDARY OUTCOMES:
prevalence of adverse events | 14 days
  At the follow-up,adverse events complained by patients will be recorded by an independent researcher，meanwhile a 8 point visual analog scale (VAS) was used to evaluate severity of adverse events.

OTHER OUTCOMES:
compliance of patients in the two groups | 14 days
  compliance was evaluated by assessing the total pills patients have taken.Compliance was defined as good when more than 80% or less than 120% of the total pills were taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hosipital, Jinan, Shandong, China